CLINICAL TRIAL: NCT05085938
Title: The Frequency of Complication and Their Causes After Gonadal Vein Embolization by Coils in Patients With Pelvic Venous Diseases
Brief Title: Complications of Gonadal Veins Embolization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Co-GAVE
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-09

CONDITIONS: Coil Embolization; Pelvic Venous Disorders; Gonadal Veins Insufficiency; Pelvic Venous Pain
Keywords: pelvic venous disorders; gonadal veins embolization; complication after coil embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gonadal veins embolisation: This group includes patients who have undergone coil embolization of gonadal vein
  Interventions: Procedure: gonadal vein embolization

INTERVENTIONS:
Procedure: gonadal vein embolization — GVE was performed under local anesthesia with 5.0-10.0 mL of 0.5% lidocaine solution with a patient under intravenous sedation. For the left GV embolization, the transfemoral approach was used, while for the right or both GV embolization, the transjugular approach was used. The 5F multipurpose angiographic catheters (Cordis; USA), standard 'moving core' J .035" guidewire, and an angled hydrophilic guidewire (Radiofocus; Terumo Corp., Japan) were used. For the GV occlusion, the pushable 0.035" standard stainless steel coils (Gianturco; William Cook, Bjæverskov, Denmark) and 0.035" coils made of Inconel with interwoven long collagen fibrils (MReye; Cook Medical Inc., Bloomington, USA) were used. The diameter of coils was 8-12 mm, and the length was 10-20 cm.

SUMMARY:
Gonadal veins embolization (GVE) with nitinol or platinum coils is widely used in the treatment of PeVD caused by the valvular incompetence of gonadal, parametrial, and uterine veins. Most authors report a high efficacy of this technique in reducing blood flow through the gonadal veins (GV) and relieving symptoms of the disease. In the Society for Vascular Surgery (SVS) and American Venous Forum (AVF) guidelines, GVE is considered the standard of treatment for PeVD with a grade of recommendation 2B, due to the moderate quality of evidence. Moreover, other studies report about wide variability in the GVE outcomes, in terms of pelvic venous pain (PVP) elimination, persistence or intensification of pain after GVE, and coil migrations and protrusions. It is known that 6% to 32% of patients do not achieve significant pain relief after the procedure. The most studies of GVE in the treatment of PeVD are characterized by only a statement of the fact of any complication without investigating the causes of its development. At the same time, it is well known that it is a thorough study of complications that makes it possible to avoid failures in the future, to improve the therapeutic technique, or to abandon its use altogether.

In this study, it is planned to conduct a retrospective analysis of patients' database, who have undergone gonadal veins embolization with nitinol coils.

DETAILED DESCRIPTION:
The aim of this study is to describe and study all side-effects and complications following embolization of gonadal veins.

This retrospective cohort study included 150 patients with PeVD who were treated by gonadal veins coil embolisation at the Savelyev University Surgical Clinic of the Pirogov Russian National Research Medical University in the period from 2000 to 2020. Patient informed consent was not required due to the retrospective nature of this study.

Inclusion criteria: the presence of symptoms and signs of PeVD (pelvic venous pain, dyspareunia, discomfort/heaviness in the hypogastric region, vulvar varicosities); reflux in the gonadal, parametrial, uterine veins according to duplex ultrasound and ovarian venography; and gonadal veins coil embolization.

Exclusion criteria: the presence of nutcracker and May-Thurner syndromes, confirmed by multiplanar renal and pelvic venography; open, endoscopic, or hybrid interventions on the gonadal and iliac veins or pelvic organs.

The diagnosis of PeVD was verified by transvaginal and transabdominal DUS, multiplanar computed tomographic venography, ovarian venography.

All patients who have undergone embolization of gonadal veins with coils were collected in a special database. The data includes parameters that can provoke complications, such as weight, duration of surgery and hospitalization, pain level before and after procedures, and others.

Gonadal vein embolization with coils:

GVE was performed under local anesthesia with 5.0-10.0 mL of 0.5% lidocaine solution with a patient under intravenous sedation. For the left GV embolization, the transfemoral approach was used, while for the right or both GV embolization, the transjugular approach was used. The vein puncture was performed under ultrasound guidance. The 5F multipurpose angiographic catheters (Cordis; USA), standard 'moving core' J .035" guidewire, and an angled hydrophilic guidewire (Radiofocus; Terumo Corp., Japan) were used. For the GV occlusion, the pushable 0.035" standard stainless steel coils (Gianturco; William Cook, Bjæverskov, Denmark) and 0.035" coils made of Inconel with interwoven long collagen fibrils (MReye; Cook Medical Inc., Bloomington, USA) were used. The diameter of coils was 8-12 mm, and the length was 10-20 cm. When selecting the coil size, the principle of 20% coil oversizing relative to the GV diameter was used in order to avoid coil migration in the conductive veins and pulmonary artery. After embolization, the control ovarian venography was performed.

Assessment of the gonadal vein embolization complications:

Complications of GVE were graded according to the Society for Interventional Radiology (SIR) Adverse Event Classification System as follows: A - No therapy, no consequences; B - Nominal therapy, no consequence; includes overnight admission for observation only; C - Requires therapy, minor hospitalization (< 48 h); D - Requires major therapy, unplanned increase in level of care, prolonged hospitalization (> 48 h); E - Permanent adverse sequelae; F - Death. Minor complications include classes A and B, and major complications include classes C to F.

Complications of gonadal vein embolization with coils included:

* Hematoma / bleeding at the access point;
* Thrombosis of non-targeted pelvic veins (parametric, uterine, internal iliac veins);
* Postembolization syndrome;
* Protrusion of coils;
* Migration of coils;
* Allergic reactions to contrast agent or nickel. Complications of gonadal vein embolization with coils were assessed within 1-30 days and 12 month after procedure.

Primary Outcome Measure:

Change in the diameter of the pelvic veins

* The diameter of the pelvic veins was measured using duplex ultrasound. [Time Frame: At baseline and 1-12 months after pelvic vein intervention.]
* Change in the duration of pelvic venous reflux Pelvic venous reflux was measured using duplex ultrasound. Reflux duration of more than 1 s was considered pathological.

[Time Frame: At baseline and 1-12 months after pelvic vein intervention.]

• Postprocedural pain The visual analogue scale is a line 10 cm long. Each centimeter corresponds to 1 point: 0 points - no pain, 10 points - maximum pain. Higher scores on the scale correspond to poorer results.

[Time Frame: 1 day, 5 days, 1 and 12 months after the intervention on the pelvic veins.] • Pelvic vein thrombosis Pelvic vein thrombosis was detected using duplex ultrasound. [Time Frame: 1 and 5 days after the intervention on the pelvic veins]

Other Pre-specified Outcome Measures:

• Complications of anesthesia Hematoma, vascular damage, pulmonary complications. [Time Frame: 1 and 5 days after the intervention on the pelvic veins]

ELIGIBILITY:
Inclusion Criteria:

* the presence of symptoms and signs of PeVD (pelvic venous pain, dyspareunia, discomfort/heaviness in the hypogastric region, vulvar varicosities);
* reflux in the gonadal, parametrial, uterine veins according to duplex ultrasound and ovarian venography;
* gonadal veins embolization with coils.

Exclusion Criteria:

* the presence of nutcracker and May-Thurner syndromes, confirmed by multiplanar renal and pelvic venography;
* open, endoscopic, or hybrid interventions on the gonadal and iliac veins or pelvic organs.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Cohort includes 150 women who have undergone gonadal vein embolisation or endoscopic resection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in the diameter of the pelvic veins | At baseline and 1-12 months after pelvic vein intervention
  The diameter of the pelvic veins was measured using duplex ultrasound
Change in the duration of pelvic venous reflux | At baseline and 1-12 months after pelvic vein intervention
  Pelvic venous reflux was measured using duplex ultrasound. Reflux duration of more than 1 s was considered pathological
Postprocedural pain | 1 day, 5 days, 1 and 12 months after the intervention on the pelvic veins
  The visual analogue scale is a line 10 cm long. Each centimeter corresponds to 1 point: 0 points - no pain, 10 points - maximum pain. Higher scores on the scale correspond to poorer results.
Pelvic vein thrombosis | 1 and 5 days after the intervention on the pelvic veins
  Thrombosis of non-targeted pelvic veins (parametric, uterine, internal iliac veins). Pelvic vein thrombosis was detected using duplex ultrasound

SECONDARY OUTCOMES:
Hemorrhagic complications | 1 and 5 days after the intervention on the pelvic veins
  Hematoma or bleeding at the access poin
Other complications after embolisation | 1 day, 5 days, 1 and 12 months after coil embolization
  Protrusion or migration of coils
Allergic reactions | 1 day, 5 days, 1 and 12 months after coil embolization
  Allergic reactions to contrast agent or nickel after procedure.

OTHER OUTCOMES:
Complications of anesthesia | 1 and 5 days after the intervention on the pelvic veins
  Hematoma, vascular damage, pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gavrilov SG, Krasavin GV, Mishakina NY, Efremova OI, Zolotukhin IA. The Effect of Venoactive Drug Therapy on the Development and Severity of Post-Embolization Syndrome in Endovascular Interventions on the Gonadal Veins. J Pers Med. 2021 Jun 7;11(6):521. doi: 10.3390/jpm11060521. PMID 34200127
- [Background] Gavrilov SG, Krasavin GV, Mishakina NY, Kirsanov KV. Postembolization syndrome in endovascular interventions on the gonadal veins. J Vasc Surg Venous Lymphat Disord. 2021 May;9(3):697-702. doi: 10.1016/j.jvsv.2020.09.003. Epub 2020 Sep 12. PMID 32932000
- [Background] Gavrilov SG, Sazhin A, Krasavin G, Moskalenko E, Mishakina N. Comparative analysis of the efficacy and safety of endovascular and endoscopic interventions on the gonadal veins in the treatment of pelvic congestion syndrome. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):178-186. doi: 10.1016/j.jvsv.2020.05.013. Epub 2020 May 25. PMID 32464289